CLINICAL TRIAL: NCT07367555
Title: Effect Of Sodium Glucose Co-Transporter-2 (SGLT-2) Inhibitors on Body Mass Index After 3 Months of Use in Diabetic Patients"
Brief Title: Effect Of Sodium Glucose Co-Transporter-2 (SGLT-2) Inhibitors on Body Mass Index After 3 Months of Use in Diabetic Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ariba Shafiq (Other)
Responsible Party: Sponsor-Investigator, Ariba Shafiq, Principal Investigator, Combined Military Hospital Multan
Organization: Combined Military Hospital Multan (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14
Record Dates: First submitted 2026-01-18; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Diabete Mellitus
Keywords: Body Mass Index; Glycemic Index; Sodium Glucose Co-transporter-2 Inhibitors
MeSH Terms: conditions — Diabetes Mellitus | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A participants with Type II Diabetes Mellitus (Experimental): Randomly 180 Individuals with diagnosed type 2 Diabetes Mellitus were allocated group A. These individuals were prescribed oral 100 gram Empagliflozin tablet along with diet plan and exercise. All individuals were followed-up in OPD for 3 months. After 3 months, individuals were assessed again for height, weight, and BMI. Changes in weight and BMI were calculated.
  Interventions: Drug: Oral 100 gram Empagliflozin tablet along with diet plan and exercise
- Group B participants with Type II Diabetes Mellitus (Active Comparator): Randomly 180 Individuals with diagnosed type 2 Diabetes Mellitus were allocated group A. These individuals were prescribed oral 100 gram Empagliflozin tablet along with diet plan and exercise. All individuals were followed-up in OPD for 3 months. After 3 months, individuals were assessed again for height, weight, and BMI. Changes in weight and BMI were calculated.
  Interventions: Other: Diet plan and exercise

INTERVENTIONS:
Drug: Oral 100 gram Empagliflozin tablet along with diet plan and exercise — oral 100 gram Empagliflozin tablet along with diet plan and exercise
  Arms: Group A participants with Type II Diabetes Mellitus
Other: Diet plan and exercise — Only Life style modification was advised. Changes in BMI were assessed.
  Arms: Group B participants with Type II Diabetes Mellitus

SUMMARY:
Total of 360 participants were enrolled and prescribed oral 200 mg SGLT-2 tablet. All participants were followed-up for about three months. Body mass index was measured before and after three months and mean change in BMI was assessed.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with type II diabetes mellitus ( blood sugar level (random) at presentation was above 186 mg/dl and HbA1c was more than 6.5% on laboratory investigations)

Exclusion Criteria:

* Individuals already taking trail drug or any other anti-glycemic drug or insulin for >6 months

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Weight | 03 Months
  Weight is measured in Kilograms

SECONDARY OUTCOMES:
Height | 03 months
  Height is measured in meters

CONTACTS AND LOCATIONS:
Overall Officials: Professor Dr Khalid Mehmood Raja, MBBS FCPS, Study Director — CMH Multan
Locations (1):
- CMH Multan, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No